CLINICAL TRIAL: NCT01202747
Title: Pilot Study for Evaluation of LipiFlow Screening Methods
Brief Title: Evaluation of Screening Methods for Treatment of Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TearScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LF002
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-11

CONDITIONS: Chalazion; Dry Eye Syndromes
MeSH Terms: conditions — Chalazion; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LipiFlow Treatment (Experimental): Treatment with LipiFlow device
  Interventions: Device: LipiFlow System

INTERVENTIONS:
Device: LipiFlow System — In-office treatment for meibomian gland dysfunction

SUMMARY:
The objective is to evaluate the feasibility of using additional screening methods to optimize effectiveness outcomes with the LipiFlow System for application of heat and pressure therapy in adult patients with chronic cystic conditions of the eyelids, including meibomian gland dysfunction, also known as evaporative dry eye or lipid deficiency dry eye, and chalazia. The screening methods include diagnostic expression of the meibomian glands and interferometry assessment of the tear film.

ELIGIBILITY:
Inclusion Criteria:

* Meibomian gland dysfunction
* Dry Eye symptoms

Exclusion Criteria:

* Ocular surgery, ocular injury or ocular Herpes infection within past 3 months
* Active ocular infection
* Active ocular inflammation or recurrent inflammation within past 3 months
* Moderate to severe allergic conjunctivitis
* Severe eyelid inflammation
* Eyelid abnormalities that affect lid function
* Ocular surface abnormalities that may compromise corneal integrity
* Systemic disease conditions or medications that cause dry eye
* Use of other treatments for meibomian gland dysfunction or dry eye
* Pregnant or nursing women
* Participation in another ophthalmic clinical trial within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Stevens, OD, Study Director — TearScience
Locations (3):
- United States (3):
  - Hoffman Estates, Illinois
  - Boston, Massachusetts
  - Winchester, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 subjects (100 eyes) were enrolled at 3 investigational sites between 10/03/2010 and 11/15/2010.
Period: Overall Study
Arm/Group | LipiFlow Treatment
Started | 50
Completed | 49 (One subject did not return for the 4 Week visit due to inconvenience.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | LipiFlow Treatment
Number analyzed (Participants) | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 49.8 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Association Between Screening Methods (Meibomian Gland Expression) and Treatment Effectiveness Outcomes (Total Meibomian Gland Score)
Description: Analysis of association between Baseline Meibomian Gland Expression Score and Total Meibomian Gland Score at 4 Weeks. Success was defined by demonstration of a statistically significant (p<0.05) association between the screening method and outcome.
  Meibomian gland expression sum scores range from 0 to 60 with a higher score reflecting less meibomian gland dysfunction. Total meibomian gland scores range from 0 to 45 with a higher score reflecting less meibomian gland dysfunction.
Time Frame: Baseline and 4 Weeks
Population: Results presented are for the Intent to Treat population.
Measure: Number; unit: Correlation coefficient
Arm/Group | LipiFlow Treatment
Number analyzed (Participants) | 50
Correlation coefficient | 0.4816
Statistical Analysis 1: Comparison: LipiFlow Treatment; Test type: Superiority or Other; p = 0.0005, Regression, Linear — p<0.05 considered statistically significant

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | LipiFlow Treatment
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No